CLINICAL TRIAL: NCT02495766
Title: Treatment of Autologous Mesenchymal Stem Cells Derived From Bone Marrow as a Potential Therapeutic Strategy for the Treatment of Multiple Sclerosis
Brief Title: Autologous Mesenchymal Stromal Cells for Multiple Sclerosis
Acronym: EMMES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Vall d'Hebron Research Institute (VHIR) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XCEL-MS-02
Record Dates: First submitted 2015-06-03; First posted 2015-07-13 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
Keywords: Multiple sclerosis; Bone marrow mesenchymal stromal cells; Stem cells; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A: XCEL-MC-ALPHA/Placebo (Experimental): Single infusion of cryopreserved bone-marrow adult mesenchymal stromal cells followed by placebo infusion at month 6.
  Interventions: Drug: XCEL-MC-ALPHA; Drug: Placebo
- Treatment B: Placebo/XCEL-MC-ALPHA (Experimental): Single infusion of placebo followed by cryopreserved bone-marrow adult mesenchymal stromal cells infusion at month 6.
  Interventions: Drug: XCEL-MC-ALPHA; Drug: Placebo

INTERVENTIONS:
Drug: XCEL-MC-ALPHA — Single infusion
  Other Names: Bone-marrow mesenchymal stromal cells
Drug: Placebo — Single infusion

SUMMARY:
This study evaluates the effect of cryopreserved autologous adult bone-marrow mesenchymal stromal cells (BM-MSC) in patients with active multiple sclerosis, compared to placebo.

Patients will be allocated to one of the 2 treatment arms (BM-MSC or placebo)and at month 6, the treatment will be crossed to receive the other product. The objective is to assess the safety of a single infusion BM-MSC, and to explore its efficacy in these patients.

Patients will be evaluated at month 12 and will be followed-up for a total of 3 years.

DETAILED DESCRIPTION:
To date, there is no effective therapy to cure multiple sclerosis (MS). Immunomodulatory therapies are useful in reducing the frequency of inflammatory processes (relapses) but don't delay significantly the progression of the disease, prevent long term disability or induce the repair of damaged tissue. This proposal contemplates the use of adult autologous bone marrow mesenchymal stromal cells (BM-MSC) as an alternative therapeutic strategy to treat patients with active MS. This is a randomized, double blind, crossover clinical trial in which 8 patients with active forms of MS and moderate disability will enter the trial with the primary objective of assessing the safety and tolerability of a single intravenous infusion of BM-MSC. Secondary objectives are to assess the efficacy by gadolinium enhancing lesions though magnetic resonance imaging, neurophysiological effects and immunological effects. Once randomized, patients will undergo BM extraction and once confirmed the availability of the needed dose, they will be randomized to one of the 2 treatment arms (BM-MSC named XCEL-MC-ALPHA, or placebo). XCEL-MC-ALPHA will be cryopreserved for all patients regardless the allocated arm. At month 6, the treatment will be crossed. Patients will be evaluated at month 12 and will be followed-up for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years of age
* Patients with MS
* Relapsing-remitting or secondary progressive MS
* Patients to whom are not indicated or are not in a position to initiate treatment with disease-modifying drugs
* Expanded Disability Status Scale (EDDS) score <6.5
* Nine T2 lesions at least
* Active multiple sclerosis as defined either by 1 outbreak in the last year or at least one Gadolinium-enhancing lesion in the last 6 months
* Signed informed consent form

Exclusion Criteria:

* Interferon beta or glatiramer acetate 3 months prior the screening
* Natalizumab or fingolimod in the 6 months prior the screening
* Mitoxantrone, cyclophosphamide or other immunosuppressive therapy at any time
* Has received an experimental treatment within 3 months prior the screening
* MS outbreak within the 4 weeks prior the randomization
* Serum creatinine> 2.0 mg/dl
* Infectious disease active or uncontrolled
* Fertile patients who are not using a suitable method of contraception
* Pregnant or lactating woman
* Immunodeficiency
* Positive serology to HIV, Hepatitis B, Hepatitis C or syphilis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | 12 months
  Safety profile

SECONDARY OUTCOMES:
Cumulative number of MRI Gd-enhancing lesions | 12 months
  Imaging procedure
Multiple Sclerosis Outbreaks | 12 months
  Medical assessment
Expanded Disability Status Scale (EDDS) score | 12 months
  Quantification of disability
Cumulative number of lesions visualized on T2 sequence | 12 months
  Imaging procedure

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Montalban, MD, PhD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Vall Hebron, Barcelona, Spain

REFERENCES:
- See also: Blood and Tissue Bank of Catalonia — http://www.bancsang.net
- See also: Multiple Sclerosis center of Catalonia — http://www.cem-cat.org/
- See also: Vall d'Hebron Research Institute — http://www.vhir.org